CLINICAL TRIAL: NCT05943080
Title: Comparison of Adductor Canal Block Combined With IPACK Block and Adductor Canal Block Combined With PCI for Postoperative Analgesia and Function Recovery Following Total Knee Arthroplasty:A Prospective, Double-Blind, Randomized Controlled Study
Brief Title: Comparison of IPACK Block and PCI for Postoperative Analgesia and Function Recovery Following Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet Fevzi Cakmak, assistant proffesor, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-12/86
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Total Knee ArthroplastyKnee Pain, Functionality
Keywords: Total Knee Arthroplasty,Knee Pain, Functionality after tka, Posterior knee analgesia
MeSH Terms: interventions — Bupivacaine; Epinephrine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: This study was designed as blinded, randomized and controlled.the person who evaluates the patients before and after the treatment is blind.In other words,the person evaluating the patients and the person giving the treatment are different.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PCI + ACB Group (Experimental): Firstly, perioperative application is performed in the anatomical space between the posterior capsule and the popliteal artery before implantation. In the application, a 22G 10 cm needle is used in the form of 20 ml 0.25% bupivacaine + 2.0 μg/mL of epinephrine.For the adductor canal block, which will be applied by the anesthesiologist at the end of the operation, first of all, the femoral artery and nerve in the inguinal region are visualized while the patient is in the supine position, accompanied by ultrasonography. Afterwards, the artery is followed distally and the adductor canal and the femoralarter inside it and the nerve are visualized. At the level just below the sartorius muscle, a simultaneous needle is visualized by ultrasonography and 7m of 0.5%bupivacaine + 8ml of 0.9% saline solution is injected into the adductor canal. Appropriate drug distribution is confirmed by ultrasonography and the procedure is terminated.
  Interventions: Drug: PCI (0.25% marcaine+ 2.0 μg/mL of adrenaline + %0.9 saline)
- IPACK block + ACB Group (Experimental): First of all, for the adductor canal block, which will be applied by the anesthesiologist at the end of the operation, the femoral artery and nerve in the inguinal region are visualized by ultrasonography while the patient is in the supine position. Afterwards, the artery is followed distally and the adductor canal and the femoral arter inside it and the nerve are visualized. At the level just below the sartorius muscle, a simultaneous needle is visualized by ultrasonography and 7m of 0.5%bupivacaine + 8ml of 0.9% saline solution is injected into the adductor canal. Appropriate drug distribution is confirmed by ultrasonography and the procedure is terminated. then ACB is performed with the help of USG in the anatomical space between the posterior capsule and the popliteal artery. In practice, a 22G 10 cm needle is used in the form of 20 ml 0.25% bupivacaine + 2.0 μg/mL of epinephrine.
  Interventions: Drug: IPACK(0.25% marcaine+ 2.0 μg/mL of adrenaline + %0.9 saline); Drug: ACB ( 0.25% marcaine + %0.9 saline)
- ACB Group (control) (Other): At the end of the operation by the anesthesiologist only adductor canal block is applied, while the patient is in the supine position, the femoral artery and nerve are visualized in the inguinal region under ultrasound guidance. Afterwards, the artery is followed distally and the adductor canal and the femoralarter inside it and the nerve are visualized. At the level just below the sartorius muscle, a simultaneous needle is visualized by ultrasonography and 7m of 0.5%bupivacaine + 8ml of 0.9% saline solution is injected into the adductor canal. Appropriate drug distribution is confirmed by ultrasonography and the procedure is terminated.
  VAS values and opioid consumption will be recorded as the primary outcome of the patients who are taken to the service after the surgical procedure performed under spinal anesthesia without the use of a tourniquet. Post-operative 3. Hour-12. Hour -24. Hours -48th hour and 72nd hour.
  Interventions: Drug: ACB ( 0.25% marcaine + %0.9 saline)

INTERVENTIONS:
Drug: PCI (0.25% marcaine+ 2.0 μg/mL of adrenaline + %0.9 saline) — The application is made into the anatomical space between the posterior capsule and the popliteal artery before implantation.
  Arms: PCI + ACB Group
Drug: IPACK(0.25% marcaine+ 2.0 μg/mL of adrenaline + %0.9 saline) — It is applied to the anatomical space between the posterior capsule and the popliteal artery with the help of USG.
  Arms: IPACK block + ACB Group
Drug: ACB ( 0.25% marcaine + %0.9 saline) — It is inserted into the adductor canal by simultaneous imaging of the needle, accompanied by ultrasonography, from the level just below the sartorius muscle.
  Arms: ACB Group (control); IPACK block + ACB Group

SUMMARY:
It was planned to determine the most effective single and/or combined use in daily use by evaluating the effect on pain control and functional status by combining the posterior capsuler infiltration (PCI) and interspace between the popliteal artery and the capsule of the posterior knee(IPACK block) performed during total knee replacement surgery with the adductor canal block method.

In the randomized controlled study:

Group 1; By determining the anatomical landmarks to be applied by the intraoperative surgeon, PCI + Adductor canal block (ACB) without any additional imaging, Group 2; IPACK+ACB applied by the anesthesiologist with the help of post-operative USG, In Group 3, there are 3 groups in which only ACB application is made. VAS values and opioid consumption of the groups will be recorded as the primary outcome after the surgery.

As a secondary outcome, the 1st day rehabilitation initiation times and endurance of the patients With 1.2. and on Day 3 joint ranges of motion will be recorded.

DETAILED DESCRIPTION:
Patients with end-stage knee osteoarthritis who were examined in our study institution and who could not respond to conservative treatment and who accepted total knee replacement (TDP) surgery will be included.

Patients will be divided into three groups by randomization: Preoperative range of motion and pain scores (VAS) of the patients will be recorded in the service examination room. By determining the anatomical landmarks to be applied by the intraoperative surgeon, they will be asked to choose one of the 3 groups in which PCI + ACB , group 2; ACB + IPACK applied by the anesthesiologist with the help of Post-operative USg, and group 3, in which only ACB application will be made, and this choice will not be known by the patient.

PCI; Perioperative application is performed in the anatomical space between the posterior capsule and the popliteal artery before implantation. In the application, a 22G 10 cm needle is used in the form of 20 ml 0.25% bupivacaine + 2.0 μg/mL of epinephrine.

IPACK: Following the closure of the wound in the postoperative period, the application is made into the anatomical space between the posterior capsule and the popliteal artery with the help of USG. In the application, 20 ml 0.25% bupivacaine + 2.0 μg/mL of epinephrine is used with a 22G 10 cm needle.

ACB: For the adductor canal block, which will be applied by the anesthesiologist at the end of the operation, the femoral artery and nerve are visualized in the inguinal region with ultrasonography while the patient is in the supine position. Afterwards, the artery is followed distally and the adductor canal and the femoralarter inside it and the nerve are visualized. At the level just below the sartorius muscle, a simultaneous needle is visualized by ultrasonography and 7m of 0.5%bupivacaine + 8ml of 0.9% saline solution is injected into the adductor canal. Appropriate drug distribution is confirmed by ultrasonography and the procedure is terminated.

VAS values and opioid consumption will be recorded as the primary outcome of the patients who are taken to the service after the surgical procedure performed under spinal anesthesia without the use of a tourniquet. Post-operative 3. Hour-12. Hour -24. Hour -48th hour and 72th hour VAS will be recorded. The total opioid consumption on the 1st, 2nd and 3rd days, when the patient needs analgesics (opioids) in the first postoperative hour will be noted.

As the Secondary Outcome, the patients' 1st day rehabilitation initiation times and their endurance are measured in 1.2. and on Day 3 joint ranges of motion will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Performing total knee joint arthroplasty due to stage 4 gonarthrosis Agree to participate in the study Having signed the informed consent form

Exclusion Criteria:

* Presence of malignancy, infection, rheumatological disease Same side has had previous surgery Known psychiatric and/or neurological diseases Expenses due to any medication or substance use

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | [Time Frame: 1 day before surgery]
  Evaluation of Pain; Visual analog scale (VAS) was used for pain assessment. VAS is in the form of a 10-point Likert scale. Patients are asked to indicate the level of pain, with 0 points as no pain, 5 points as moderate pain, and 10 points as unbearable pain. Increased scores indicate higher pain level.
Pain Intensity | [Time Frame: 3th hour after surgery]
  Evaluation of Pain; Visual analog scale (VAS) was used for pain assessment. VAS is in the form of a 10-point Likert scale. Patients are asked to indicate the level of pain, with 0 points as no pain, 5 points as moderate pain, and 10 points as unbearable pain. Increased scores indicate higher pain level.
Pain Intensity | [Time Frame: 8th hour after surgery]
  Evaluation of Pain; Visual analog scale (VAS) was used for pain assessment. VAS is in the form of a 10-point Likert scale. Patients are asked to indicate the level of pain, with 0 points as no pain, 5 points as moderate pain, and 10 points as unbearable pain. Increased scores indicate higher pain level.
Pain Intensity | [Time Frame: 12th hour after surgery]
  Evaluation of Pain; Visual analog scale (VAS) was used for pain assessment. VAS is in the form of a 10-point Likert scale. Patients are asked to indicate the level of pain, with 0 points as no pain, 5 points as moderate pain, and 10 points as unbearable pain. Increased scores indicate higher pain level.
Pain Intensity | [Time Frame: 24th hour after surgery]
  Evaluation of Pain; Visual analog scale (VAS) was used for pain assessment. VAS is in the form of a 10-point Likert scale. Patients are asked to indicate the level of pain, with 0 points as no pain, 5 points as moderate pain, and 10 points as unbearable pain. Increased scores indicate higher pain level.
Pain Intensity | [Time Frame: 48th hour after surgery]
  Evaluation of Pain; Visual analog scale (VAS) was used for pain assessment. VAS is in the form of a 10-point Likert scale. Patients are asked to indicate the level of pain, with 0 points as no pain, 5 points as moderate pain, and 10 points as unbearable pain. Increased scores indicate higher pain level.
Pain Intensity | [Time Frame: 72th hour after surgery]
  Evaluation of Pain; Visual analog scale (VAS) was used for pain assessment. VAS is in the form of a 10-point Likert scale. Patients are asked to indicate the level of pain, with 0 points as no pain, 5 points as moderate pain, and 10 points as unbearable pain. Increased scores indicate higher pain level.
opioid usage | first hour of use
  usage vanalgesics (opioids) in the first postoperative hour
opioid comsuption | [Time Frame: 24th hour after surgery]
  opioid consumption after surgery
opioid comsuption | [Time Frame: 48th hour after surgery]
  opioid consumption after surgery
opioid comsuption | [Time Frame: 72th hour after surgery]
  opioid consumption after surgery

SECONDARY OUTCOMES:
Measuring knee Joint Range of Motion | [Time Frame: 1 day before surgery]
  Knee joint range of motion (ROM) measurement with goniometer is the most commonly used method that provides objective evaluation and error-free measurement in clinical practice. In our study, knee ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Measuring knee Joint Range of Motion | [Time Frame: 1 days after before surgery]
  Knee joint range of motion (ROM) measurement with goniometer is the most commonly used method that provides objective evaluation and error-free measurement in clinical practice. In our study, knee ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Measuring knee Joint Range of Motion | [Time Frame: 3 days after surgery]
  Knee joint range of motion (ROM) measurement with goniometer is the most commonly used method that provides objective evaluation and error-free measurement in clinical practice. In our study, knee ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Measuring knee Joint Range of Motion | [Time Frame: 10 days after surgery]
  Knee joint range of motion (ROM) measurement with goniometer is the most commonly used method that provides objective evaluation and error-free measurement in clinical practice. In our study, knee ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahievran university, Kirşehi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beswick AD, Wylde V, Gooberman-Hill R, Blom A, Dieppe P. What proportion of patients report long-term pain after total hip or knee replacement for osteoarthritis? A systematic review of prospective studies in unselected patients. BMJ Open. 2012 Feb 22;2(1):e000435. doi: 10.1136/bmjopen-2011-000435. Print 2012. PMID 22357571
- [Result] Niesen AD, Harris DJ, Johnson CS, Stoike DE, Smith HM, Jacob AK, Amundson AW, Pawlina W, Martin DP. Interspace between Popliteal Artery and posterior Capsule of the Knee (IPACK) Injectate Spread: A Cadaver Study. J Ultrasound Med. 2019 Mar;38(3):741-745. doi: 10.1002/jum.14761. Epub 2018 Sep 19. PMID 30232819
- [Result] Sankineani SR, Reddy ARC, Eachempati KK, Jangale A, Gurava Reddy AV. Comparison of adductor canal block and IPACK block (interspace between the popliteal artery and the capsule of the posterior knee) with adductor canal block alone after total knee arthroplasty: a prospective control trial on pain and knee function in immediate postoperative period. Eur J Orthop Surg Traumatol. 2018 Oct;28(7):1391-1395. doi: 10.1007/s00590-018-2218-7. Epub 2018 May 2. PMID 29721648